CLINICAL TRIAL: NCT01784978
Title: Randomized ph. II Study to Explore Efficacy and Feasibility of Upfront Rotations Between SUNitinib and Everolimus vs Sequential Treatment of 1st lIne Sunitinib & 2nd Line EverolimuS Until Progression in Pats Met. Clear Cell Renal Cancer
Brief Title: Efficacy Study of Sunitinib and Everolimus (Rotational vs Sequential Arm) in Pats. With m Clear Cell Renal Cancer
Acronym: SUNRISES
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Associació per a la Recerca Oncologica, Spain (Other)
Collaborators: Novartis (Industry); Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUNRISES STUDY (CRAD001LIC34T)
Record Dates: First submitted 2012-12-11; First posted 2013-02-06 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: cancer; renal; metastatic; clear; cell; Sunitinib; Everolimus; Alternating
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Neoplasm Metastasis; Margins of Excision | interventions — Sunitinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rotational arm (Experimental): Alternating cycles of treatment with sunitinib and everolimus; repeating cycles of 24 weeks of treatment consisting of 12 weeks of sunitinib 4weeks on 2 weeks off, 50 mg pd followed by 12 weeks of everolimus 10 mg per day 11 weeks on 1 week off in patients with metastatic clear cell renal cancer.
  Interventions: Drug: Sunitinib; Drug: Everolimus
- Sequential arm (Active Comparator): The comparative arm will be the standard regimen of sunitinib (50 mg pd 4/2) until progression, followed thereafter by everolimus (10 mg per day continuously, 11/1) until progression.
  Interventions: Drug: Sunitinib; Drug: Everolimus

INTERVENTIONS:
Drug: Sunitinib — 50 mg pd
  Other Names: SUTENT
Drug: Everolimus — 10 mg pd
  Other Names: AFINITOR

SUMMARY:
The objective of this study is to assess the progression-free survival, of patients who receive rotations of sunitinib and everolimus versus patients who receive sunitinib as a first line treatment followed by everolimus when progression occurs.

DETAILED DESCRIPTION:
This is an open-label, randomized phase II study to investigate the feasibility of alternating cycles of treatment with sunitinib and everolimus compared to sequential treatment of sunitinib followed by everolimus.

The study population consists of adult patients (over 18 years old) with clear cell mRCC (Metastatic Renal Cell Cancer) who have not received prior therapy for their metastatic disease.

The purpose of the study is to determine the progression free survival, feasibility and safety profile of the experimental arm compared to standard of care.

In the experimental arm alternating treatment will consist of repeating cycles of 24 weeks of treatment consisting of 12 weeks of sunitinib 4weeks on 2 weeks off, 50 mg pd followed by 12 weeks of everolimus 10 mg per day 11 weeks on 1 week off in patients with metastatic clear cell renal cancer. The comparative arm will be the standard regimen of sunitinib (50 mg pd 4/2) until progression, followed thereafter by everolimus (10 mg per day continuously, 11/1) until progression.

ELIGIBILITY:
Inclusion Criteria:

* Renal cell carcinoma with a predominant clear cell component confirmed by histology.
* Advanced disease: metastatic AND, not suitable for resection
* Male or female, aged 18 years or older
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0 or 1
* Low or intermediate MSKCC (Memorial Sloan Kettering Cancer Center) prognostic risk score,i.e. no more than 2 of the following:

  * Karnofsky performance status (<80%)
  * Low serum hemoglobin (≤ 13 g/dL for males and ≤ 11.5 g/dL for females)
  * High corrected serum calcium (≥ 10 mg/dL)
* Target and/or non-target lesions according to RECIST 1.1 ( Response Evaluation Criteria in Solid Tumors)
* Expected survival of at least 3 months.
* No prior systemic treatment. But adjuvant treatment is ok if stopped from ≥ 24 months
* Adequate bone marrow function as shown by:
* Adequate liver function as shown by:
* Adequate renal function as shown by serum creatinine ≤ 1.5 x ULN (upper limit of normal)
* Left ventricular ejection fraction ≥55% on gated cardiac blood pool scan, or normal left ventricular function and fractional shortening on echocardiogram (according to institutional limits).
* SBP (systolic blood pressure) ≤140mmHg and DBP (diastolic blood pressure)

  * 90mmHg (it is acceptable to initiate antihypertensive treatment prior to registration to achieve these goals).
* Able to commence treatment within 7 days of registration.
* Willing and able to comply with follow-up and all other protocol requirements.
* Written informed consent

Exclusion Criteria:

* Prior treatment with VEGF-targeting agents or multi-kinase inhibitors or mTOR-targeting agents
* Active central nervous system metastases.
* Other malignancy diagnosed within the last 5 years, except the following if adequately treated: superficial squamous cell carcinoma or basal cell carcinoma of skin, superficial bladder cancer (T1 and G1 or T1 and G2), stage 1 cervical cancer.
* Treatment with an investigational agent in the last 4 w.
* Known to be HIV positive.
* Evidence of chronic hepatitis due to hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Clinically significant heart disease (NYHA Class III or IV)
* History of hypertension requiring hospitalization.
* Other serious illnesses,
* Immunotherapy or chemotherapy in the last 4 w (6 weeks for nitrosoureas)
* Major surgery in the last 4 w, or planned in the next 6 w
* Radiation therapy in the last 2 w, or planned in the next 6 w
* NCI CTCAE (Common Toxicity Criteria for Adverse Effects) version 4.0 grade 3 or worse hemorrhage in last 4 w.
* Any of the following in the last year: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
* Ongoing cardiac dysrhythmias of NCI CTCAE version 4.0 grade ≥2, atrial fibrillation of any grade, or prolongation of the corrected QT interval (QTc) to >450 msec for males or >470 msec for females
* Uncontrolled diabetes as defined by fasting serum glucose >1.5 X ULN.
* Pregnancy,lactation. Inadequate contraception.
* Known allergy or hypersensitivity to everolimus, sunitinib or iodine.
* Medical or psychiatric condition that compromises the patient's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-02-12 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate 1 year | 12 months

SECONDARY OUTCOMES:
PFS of rotational arm versus PFS of the 2 lines in control arm | From date of randomization until the date of first documented progression assesed up to 30 months
Overall Survival | From the date of the tratment start to the date of death or the last contact for alived patients at the momment of data censored. Assesed up to 30 months
Safety Profile | From the first treatment dose until 28 days after study treatment discontinuation. Assesed up to 30 months
Objective tumor response rate per arm | From the date of first tumor response to the date of progression or start date of other cancer therapy. Assesed up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Bellmunt, MD/PhD, Principal Investigator — Associacio Per la Recerca Oncológica (APRO)
Locations (10):
- Hopital Bordeaux University, Bordeaux, France
- ALEXANDRA General Hospital of Athens, Athens, Greece
- Spain (8):
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital del Mar, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Clara Campal. Hospital Sanchinarro, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Rodriguez-Vida A, Bamias A, Esteban E, Saez MI, Lopez-Brea M, Castellano D, Caballero C, Gonzalez-Larriba JL, Calvo E, Macia S, Ravaud A, Bellmunt J. Randomised Phase II study comparing alternating cycles of sunitinib and everolimus vs standard sequential administration in first-line metastatic renal carcinoma (SUNRISES study). BJU Int. 2020 Nov;126(5):559-567. doi: 10.1111/bju.15165. Epub 2020 Aug 2. PMID 32654362